CLINICAL TRIAL: NCT02774382
Title: Rectal Bacteriotherapy, Fecal Microbiota Transplantation or Oral Vancomycin Treatment of Recurrent Clostridium Difficile Infections
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Andreas Munk Petersen, MD, PhD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJ-478
Record Dates: First submitted 2016-04-04; First posted 2016-05-17 (Estimated); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Clostridium Difficile
Keywords: Recurrence; Infection
MeSH Terms: conditions — Recurrence; Infections | interventions — Vancomycin; Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vancomycin (Active Comparator): Oral vancomycin according to number of recurrences (Danish guidelines):
  First recurrence: Capsule vancomycin 125 mg x 4 p.o. times daily for 14 days
  ≥2 recurrences:
  * capsule vancomycin 125 mg x 4 times daily p.o. for 14 days followed by
  * capsule vancomycin 125 mg x 2 times daily p.o. for 7 days followed by
  * capsule vancomycin 125 mg x 1 times daily p.o. for 7 days followed by
  * capsule vancomycin 125 mg x 1 p.o. every second day for 7 days followed by
  * capsule vancomycin 125 mg x 1 p.o. every third day for 14 days
  Interventions: Drug: Vancomycin
- Vancomycin + fecal microbiota transplantation (Experimental): Capsule vancomycin 125 mg x 4 times daily p.o. for 7-14 days followed by Fecal Microbiota Transplantation with 200 ml fecal suspension administrated with a rectal catheter.
  Interventions: Drug: Vancomycin; Drug: Fecal microbiota transplantation
- Vancomycin + rectal bacteriotherapy (Experimental): Capsule vancomycin 125 mg x 4 times daily p.o. for 7-14 days followed by Rectal bacteriotherapy with 200 ml suspension of a fixed mixture of bacterial strains administrated with a rectal catheter.
  Interventions: Drug: Vancomycin; Drug: Rectal bacteriotherapy

INTERVENTIONS:
Drug: Vancomycin — Already incl. in arm description
Drug: Fecal microbiota transplantation — Already incl. in arm description
  Arms: Vancomycin + fecal microbiota transplantation
Drug: Rectal bacteriotherapy — Already incl. in arm description
  Arms: Vancomycin + rectal bacteriotherapy

SUMMARY:
The purpose of the study is to investigate if treatment with fecal microbiota transplantation or rectal bacteriotherapy is superior to standard vancomycin in patients with recurrent Clostridium Difficile infections.

DETAILED DESCRIPTION:
Clostridium difficile infection (CDI) is the most common nosocomial infection in the western world. CDI is associated with high morbidity and mortality and is a great burden for the health care system leading Center of Disease Control and Prevention (CDC) to identify it as one of three most important/urgent threats to public health.

Despite antimicrobial treatment of CDI, 20% of the patients have recurrence of CDI. Due to a dysbiosis in the gut microbiota the antimicrobial treatment seems to be less effective.

Fecal microbiota transplantation (FMT) is an alternative treatment for recurrent CDI. Studies have shown a cure rate up to 90% in patients with recurrent CDI. One alternative to FMT is rectal bacteriotherapy (RBT) which is a standardized bacterial culture made in the laboratory consisting of 12 different bacteria. RBT has never been investigated in a clinical trial.

The project is a randomized controlled trial including 450 patients with recurrent CDI will be, after accepting participation, allocated to receive vancomycin alone or vancomycin followed by either FMT or RBT. The patients will be followed up for 180 days. Cure is defined as resolution of CDI symptoms 90 days after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Verified recurrent CDI with symptoms of CDI and microbiological verification (PCR).
* Previously treated for CDI with at least 10 days of vancomycin or metronidazole.
* Be able to read and understand Danish.

Exclusion Criteria:

* Life expectancy < 3 months.
* Allergy toward vancomycin
* Other infection in the GI tract with clinical symptoms similar to CDI.
* Other illness in the GI tract with clinical symptoms similar to CDI.
* Use of antibiotics for more than 14 days treating other infections
* Planning pregnancy, pregnancy or breast feeding.
* Severe immune suppression which makes FMT/RBT relatively contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Clinical cure of recurrent Clostridium difficile infection defined as patient-reported abscence of Clostridium difficile infection 90 days after treatment. | 90 days
  Clinical cure defined as patient-reported abscence of Clostridium difficile infection 90 days after treatment. The investigator will call the patient by telephone and fill out af digital questionnaire.

SECONDARY OUTCOMES:
Early or late recurrence of CDI after the end of treatment defined as recurrence of symptoms of CDI and a positive stool sample with Clostridium difficile (PCR). | 30 and 180 days after ended treatment
  Patient with recurrence of CDI in the follow up period will be categorized as an early recurrence if the recurrence is in the first 30 days after treatment and as a late recurrence if the recurrence is after 180 days after treatment. The investigator will call the patient by telephone and fill out af digital questionnaire and thereafter categorize the patient.
Days with diarrhea | 1, 4, 8 and 12 days after ended treatment
CDI-associated hospital admission and hospital admission of other causes in the follow-up period | 180 days after ended treatment
CDI-associated hospital outpatient contact and hospital outpatient contact of other causes in the follow-up period | 180 days after ended treatment
CDI-associated mortality and all-cause mortality | 30, 90 and 180 days after ended treatment
Compare numbers of patients with clinical cure after study treatment divided into two groups depending on numbers of recurrences of CDI. | 90 days after ended treatment
  Clinical cure is defined as patient-reported abscence of Clostridium difficile infection 90 days after treatment. The investigator will call the patient by telephone and fill out a digital questionnaire. Number of patients with clinical cure of recurrent Clostridium difficile infection will be divided into two groups according to numbers of recurrences of CDI;
  * Group 1; patients with one recurrence
  * Group 2; patients with 2 or more recurrences. The division will be done based on patient records and the questionnaire. The information will be aggregated in the digital journal unique to this trial. The numbers of patients with clinical cure in the two groups will be compared to see if one group response better to study treatment than the other.
Effect of the treatment depending on the CD strain - i.e. toxin B CDI cases, toxin B plus binary toxin CDI cases and CD027 CDI cases. | 90 days after ended treatment
  The investigator will call the patient by telephone and fill out af digital questionnaire. The lab result will give the investigator information about which strain the patient was infected with and this will be aggregated in the digital patient journal.
Effect of the treatment depending on the patients serum-level of antibodies towards toxin A and B at the time of inclusion. | 90 days after ended treatment
  At inclusion the investigator will collect a blood sample to analysis for toxin A and B antibodies. The lab result will be aggregated in the digital patient journal.
Side effects in the three treatment arms | 14 days after ended treatment
Characterisation of the gut microbiota before and after treatment with FMT/RBT in conjunction with characterisation of the donor's microbiota or the RBT bacterial mix. | 180 days after ended treatment
  Performed in a subgroup of patients.
Other antibiotic treatments associated with new recurrences of CDI | Within 180 days after ended treatment
  The investigator will call the patient by telephone and fill out af digital questionnaire. Furthermore the investigator has access to a database with all prescription drugs incl. antibiotics. These informations will be collected and aggregated in the digital patient journal unique for this study.
Evaluation of the composition of bile acids before and after treatment with FMT/RBT. | 90 days after ended treatment
  Analyzed in conjunction with the microbiota composition and the treatment effect. Performed in a subgroup of patients.
Characterisation of the CD strains by whole genome sequencing | 90 days after ended treatment
  Characterisation of the CD strains involved to determine if a potential recurrence is a true recurrence or a reinfection with another strain. Whole genome sequencing will be performed by the department of Clinical Microbiology in Hvidovre Hospital. This information will be collected by the investigator and aggregated in the digital patient journal unique for this trial.
Identification of age as a risk factor for treatment success/failure | 90 days after ended treatment
  The investigator will call the patient by telephone for information about abscence of CDI and fill out af digital questionnaire. This information and the patient's age will be aggregated in the digital patient journal.
Identifying if Charlson comorbidity index is associated to treatment success/failure. | 90 days after ended treatment
  At inclusion the patient's Charlson Comorbidity index will be calculated and put in the patient's record unique to this trial.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas M Petersen, MD PhD, Principal Investigator — Hvidovre University Hospital
Locations (2):
- Denmark (2):
  - Hvidovre Hospital, Hvidovre
  - Køge sygehus, Køge

REFERENCES:
- [Background] Kelly CP, LaMont JT. Clostridium difficile--more difficult than ever. N Engl J Med. 2008 Oct 30;359(18):1932-40. doi: 10.1056/NEJMra0707500. No abstract available. PMID 18971494
- [Background] Lessa FC, Mu Y, Bamberg WM, Beldavs ZG, Dumyati GK, Dunn JR, Farley MM, Holzbauer SM, Meek JI, Phipps EC, Wilson LE, Winston LG, Cohen JA, Limbago BM, Fridkin SK, Gerding DN, McDonald LC. Burden of Clostridium difficile infection in the United States. N Engl J Med. 2015 Feb 26;372(9):825-34. doi: 10.1056/NEJMoa1408913. PMID 25714160
- [Background] Olsen MA, Yan Y, Reske KA, Zilberberg MD, Dubberke ER. Recurrent Clostridium difficile infection is associated with increased mortality. Clin Microbiol Infect. 2015 Feb;21(2):164-70. doi: 10.1016/j.cmi.2014.08.017. Epub 2014 Oct 12. PMID 25658560
- [Background] van Nood E, Vrieze A, Nieuwdorp M, Fuentes S, Zoetendal EG, de Vos WM, Visser CE, Kuijper EJ, Bartelsman JF, Tijssen JG, Speelman P, Dijkgraaf MG, Keller JJ. Duodenal infusion of donor feces for recurrent Clostridium difficile. N Engl J Med. 2013 Jan 31;368(5):407-15. doi: 10.1056/NEJMoa1205037. Epub 2013 Jan 16. PMID 23323867
- [Background] Cammarota G, Masucci L, Ianiro G, Bibbo S, Dinoi G, Costamagna G, Sanguinetti M, Gasbarrini A. Randomised clinical trial: faecal microbiota transplantation by colonoscopy vs. vancomycin for the treatment of recurrent Clostridium difficile infection. Aliment Pharmacol Ther. 2015 May;41(9):835-43. doi: 10.1111/apt.13144. Epub 2015 Mar 1. PMID 25728808
- [Background] Tvede M, Tinggaard M, Helms M. Rectal bacteriotherapy for recurrent Clostridium difficile-associated diarrhoea: results from a case series of 55 patients in Denmark 2000-2012. Clin Microbiol Infect. 2015 Jan;21(1):48-53. doi: 10.1016/j.cmi.2014.07.003. Epub 2014 Oct 12. PMID 25636927